CLINICAL TRIAL: NCT00768534
Title: Microbiological Analysis Of Spontaneous Draining Acute Otitis Media Including Serotype Distribution Of Pneumococcal Isolates
Brief Title: Study Evaluating Microbiological Analysis of Spontaneous Draining Acute Otitis Media
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0887X1-4454; B1841014 (Other: Alias Study Number)
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Otitis Media
Keywords: Acute Otitis Media; Serotype distribution
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Middle ear fluid and anasopharyngeal swab
Oversight: Data Monitoring Committee: No

SUMMARY:
Describe the patient population and bacterial microbiology of pediatric patients presenting with spontaneous draining acute otitis media

ELIGIBILITY:
Inclusion Criteria:

Main inclusion criteria:

* Children >= 2 months and =< 5 years
* Spontaneous draining AOM =< 2 days Main

Exclusion Criteria:

exclusion criteria:

* Previous operation of the ear
* Chronic otitis media or tube placement with drainage >= 3 days
* Chronic disease/immune deficiency

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 2138 (Actual)
Dates: Start 2008-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
serotype distribution | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Dr. Andreas Busse, Tegernsee, Bavarian, Germany

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0887X1-4454&StudyName=Study%20Evaluating%20Microbiological%20Analysis%20of%20Spontaneous%20Draining%20Acute%20Otitis%20Media